CLINICAL TRIAL: NCT01775501
Title: Phase II Trial of Sorafenib in Combination With Modified FOLFOX in Patients With Advanced Hepatocellular Carcinoma
Brief Title: Sorafenib + mFOLFOX for Hepatocellular Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Goyal, Lipika, Prinicipal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-218
Record Dates: First submitted 2013-01-18; First posted 2013-01-25 (Estimated); Results first posted 2020-04-22 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Hepatocellular Cancer
Keywords: sorafenib; FOLFOX
MeSH Terms: conditions — Liver Neoplasms | interventions — Leucovorin; Fluorouracil; Oxaliplatin; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Experimental Treatment Arm (Experimental): FOLFOX (Leucovorin, Fluorouracil and Oxaliplatin) + Sorafenib Sorafenib: orally, twice daily FOLFOX: injected via portacath once every two weeks
  Interventions: Drug: Leucovorin; Drug: Fluorouracil; Drug: Oxaliplatin; Drug: Sorafenib

INTERVENTIONS:
Drug: Leucovorin — 200mg/m2 administered IV on Days 1 and 15 of a 28 day cycle. Number of Cycles: until progression or unacceptable toxicity develops.
  Other Names: Folinic acid
Drug: Fluorouracil — 5-FU continuous infusion: 2400mg/m2 total (1200mg/m2/d on day 1 and 2) to start on Day 1 and Day 15 of each 28 day cycle. Number of Cycles: until progression or unacceptable toxicity develops.
  Other Names: 5-FU
Drug: Oxaliplatin — 85 mg/m2 IV on Days 1 and 15 of each 28 day cycle. Number of Cycles: until progression or unacceptable toxicity develops.
  Other Names: Eloxatin
Drug: Sorafenib — 400mg po BID continuously for a 2 week lead-in phase and then Days 1-28 of each 28 day cycle. Number of Cycles: until progression or unacceptable toxicity develops.
  Other Names: Nexavar

SUMMARY:
This research study is a Phase II clinical trial. Phase II clinical trials test the effectiveness of an investigational combination of drugs to learn whether the drug combination works in treating a specific cancer. "Investigational" means that the modified FOLFOX and sorafenib combination is still being studied and that research doctors are trying find out more about it-such as the safest dose to use, the side effects it may cause, and if the combination is effective for treating different types of cancer. It also means that the FDA has not yet approved the modified FOLFOX and sorafenib combination that will be used in this study for liver cancer.

FOLFOX is a combination of three drugs: folinic acid (leucovorin), fluorouracil (5-FU), and oxaliplatin. The dosage amounts for some of these FDA approved drugs will be modified slightly in this study. The FOLFOX combination is approved by the FDA and is a standard treatment of colorectal cancer. However, it is not approved for the treatment of liver cancer.

Sorafenib is a new drug, which is approved under the brand name Nexavar for the treatment of liver cancer. It is also currently being tested in various other cancers. Sorafenib works by slowing down and/or stopping the development of new cancer cells and new blood vessels. By slowing down and/or stopping the growth of new blood vessels around a tumor, it is believed that sorafenib prevents or slows down the growth of tumors.

In this research study, sorafenib, the standard treatment, is being combined with modified FOLFOX, which has shown some antitumor activity in liver cancer.

DETAILED DESCRIPTION:
After agreeing to participate in this study, the patient will be asked to undergo some screening tests or procedures to find out if he/she is eligible. Many of these tests and procedures are likely to be part of regular cancer care and may be done even if it turns out that the patient does not take part in the research study. If the patient has had some of these tests or procedures recently, they may or may not have to be repeated. These tests and procedures include: a medical history, physical exam, performance status, electrocardiogram, assessment of tumor, blood tests, urine test, pregnancy test and optional research biopsy. If these tests show that the patient is eligible to participate in the research study, he/she will begin the study treatment. If the patient does not meet the eligibility criteria, he/she will not be able to participate.

If the patient takes part in this research study, he/she will be given a sorafenib study drug-dosing diary for each treatment cycle. Each treatment cycle lasts 28 days (4 weeks), during which time the patient will be taking the study drug twice daily. The diary will also include special instructions for sorafenib.

There will be a 2-week Lead-in period, in which the patient will receive sorafenib alone for the first two weeks of the study. Cycle 1 will begin once the patient receives the combination sorafenib and FOLFOX.

For FOLFOX, all three chemotherapy drugs will be injected through a central vein in the patient's chest (portacath) and will be given once every two weeks (14 days), starting on Day 15 of Cycle 1. The patient will receive oxaliplatin first as a 2-hour infusion, followed by leucovorin, and then 5-FU. The 5-FU infusion can last up to 46 hours and will be given through a small portable pump. The investigator will ask the patient to come back to the clinic on day 3 (46 hours after begin 5-FU dose) for pump discontinuance.

During all cycles the patient will have a physical exam and the patient will be asked questions about his/her general health and specific questions about any problems that he/she might be having and any medication he/she may be taking.

As part of the research study the patient will undergo research blood tests that will measure certain proteins in the blood to learn what affect the study treatment may have on you and your disease. About 1 teaspoon of blood will be drawn on Days 3 and 14 during your first two weeks of sorafenib alone, again on Days 14 and 28 post-treatment with FOLFOX-sorafenib and, if available, at the time of progression (if the patient's disease gets worse).

The patient's blood pressure will be monitored once every week for the first 6 weeks of the study (once a week during sorafenib lead-in period and Cycle 1). The investigator will asses the patient's tumor by chest, abdominal and pelvic CT or MRI scan once every 8 weeks throughout the study.

After the final dose of the study drug the investigator will ask the patient to come back to the clinic to repeat the following procedures: medical review, physical examination, blood tests, pregnancy test and tumor assessment by CT or MRI. The investigator would like to keep track of patient's medical condition for the rest of his/her life. The investigator would like to do this by calling the patient on the telephone once a year to see how the patient is doing. Keeping in touch with the patient and checking his/her condition every year helps the investigator look at the long-term effects of the research study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed advanced HCC
* Barcelona Clinic Liver Cancer stage C or stage B if you cannot tolerate or failed TACE
* No cirrhosis or Child-Pugh A cirrhosis
* Measurable lesions
* All acute toxic effects of any prior treatment have resolved to NCI-CTCAE v4.0 grade 1 or less
* Able to swallow and retain oral medication

Exclusion Criteria:

* Prior systemic regimens for HCC
* Uncontrolled hypertension
* CLIP score > 3
* ECOG PS > 1
* Clinically apparent central nervous system metastases or carcinomatous meningitis
* Pregnant or breastfeeding
* Active or clinically significant cardiac disease
* Evidence or history of bleeding diathesis or coagulopathy
* Any pulmonary hemorrhage/bleeding event of NCI-CTCAE v4.0 Grade 2 or higher within 4 weeks of enrollment
* Presence of a non-healing wound, non-healing ulcer, or bone fracture
* History of organ allograft
* Any malabsorption condition
* Medical or psychiatric condition that constitutes an unacceptable risk for participation in this trial
* Have received another investigational agent within 4 weeks of first dose of sorafenib
* Previously untreated or concurrent cancer except those treated more than 3 years ago
* History of other disease, metabolic dysfunction, physical examination finding or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that might affect the interpretation of the results of the study or render the subject at high risk from treatment complications
* QTC>500msec or history of uncontrolled angina, arrhythmias, or congestive heart failure
* Concurrent systemic and local anti-cancer therapy
* Prior use of sorafenib, oxaliplatin or 5FU
* Major surgery within 30 days
* Concurrent use of aspirin>100mg
* Therapeutic anticoagulation with vitamin K antagonists or with heparins or heparinoids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2019-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lipika Goyal, MD, Principal Investigator — MGH
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts

RESULTS

PARTICIPANT FLOW:
Groups:
- FOLFOX + Sorafenib: FOLFOX (Leucovorin, Fluorouracil and Oxaliplatin) + Sorafenib Sorafenib: orally, twice daily FOLFOX: injected via portacath once every two weeks
  Leucovorin: 200mg/m2 administered IV on Days 1 and 15 of a 28 day cycle. Number of Cycles: until progression or unacceptable toxicity develops.
  Fluorouracil: 5-FU continuous infusion: 2400mg/m2 total (1200mg/m2/d on day 1 and 2) to start on Day 1 and Day 15 of each 28 day cycle. Number of Cycles: until progression or unacceptable toxicity develops.
  Oxaliplatin: 85 mg/m2 IV on Days 1 and 15 of each 28 day cycle. Number of Cycles: until progression or unacceptable toxicity develops.
  Sorafenib: 400mg po BID continuously for a 2 week lead-in phase and then Days 1-28 of each 28 day cycle. Number of Cycles: until progression or unacceptable toxicity develops.
Period: Overall Study
Arm/Group | FOLFOX + Sorafenib
Started | 40
Completed | 39
Not Completed | 1
Not completed — Discontinued prior to treatment | 1

BASELINE CHARACTERISTICS:
Arm/Group | FOLFOX + Sorafenib
Number analyzed (Participants) | 40
Age, Continuous [Median (Full Range); unit: years] | 65 [29 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 34
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 35
  Black | 1
  Asian | 1
  Not Reported | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Time to Progression
Description: The median amount of time from the time of registration until disease progression. Disease progression was assessed using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
  Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
Time Frame: The amount of time from registration until disease progression or death, median duration 7.7 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | FOLFOX + Sorafenib
Number analyzed (Participants) | 40
Months | 7.7 [4.4 to 8.9]

2. Secondary Outcome: Number of Patients Experiencing Adverse Events
Description: To evaluate the tolerability and toxicities of FOLFOX-S regimen in this population of patients.
Time Frame: From the start of treatment until 30 days after the end of treatment, median duration of 10.7 months
Measure: Count of Participants; unit: Participants
Arm/Group | FOLFOX + Sorafenib
Number analyzed (Participants) | 40
Participants | 40

3. Secondary Outcome: Overall Response Rate
Description: Overall response rate is the number of participants that achieved either a complete or partial response according to RECIST 1.1 criteria.
  * Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  * Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | FOLFOX + Sorafenib
Number analyzed (Participants) | 39
Participants | 7

4. Secondary Outcome: Median Progression Free Survival
Description: The median duration of time from the start of treatment until disease progression or death
Time Frame: From the start of treatment until disease progression or death, median duration of 232 days
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | FOLFOX + Sorafenib
Number analyzed (Participants) | 40
Days | 232 [118 to 306]

5. Secondary Outcome: Median Overall Survival
Description: The duration of time from study registration until death.
Time Frame: From registration until death, median duration of 15.1 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | FOLFOX + Sorafenib
Number analyzed (Participants) | 40
Months | 15.1 [7.9 to 16.9]

6. Secondary Outcome: Duration of Response
Description: The median amount of time from achieving a response (partial or complete) until disease progression, death, or loss to follow-up.
Time Frame: From the time of treatment response until death or disease progression (median duration 172 days)
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | FOLFOX + Sorafenib
Number analyzed (Participants) | 40
Days | 172 [112 to NA] — Upper limit of the confidence interval is not estimable due to an insufficient number of participants with events

ADVERSE EVENTS:
Time Frame: From the start of treatment until 30 days after the end of treatment, median duration of 10.7 months
Arm/Group | FOLFOX + Sorafenib
All-Cause Mortality (participants affected / at risk) | 2/40
Serious Adverse Events (participants affected / at risk) | 32/40
Other Adverse Events (participants affected / at risk) | 40/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FOLFOX + Sorafenib (N=40)
Alanine aminotransferase increased (Investigations) | 6 (6)
Alkaline phosphatase increased (Investigations) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 3 (4)
Aspartate aminotransferase increased (Investigations) | 9 (12)
Bleeding (Epistaxis, Hematuria, Hematoma, Hemorrhoidal hemorrhage, Rectal hemorrhage) (Gastrointestinal disorders) | 1 (1)
Blood bilirubin increased (Investigations) | 4 (4)
Diaphoresis (Skin and subcutaneous tissue disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 4 (4)
Fatigue (General disorders) | 3 (3)
Fever (General disorders) | 1 (1)
Flushing (Vascular disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 2 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 13 (25)
Lipase increased (Investigations) | 9 (11)
Lymphocyte count decreased (Investigations) | 7 (12)
Mouth Sores (Gastrointestinal disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 3 (4)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 3 (4)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Platelet count decreased (Investigations) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (2)
Serum amylase increased (Investigations) | 2 (2)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FOLFOX + Sorafenib (N=40)
Abdominal distension (Gastrointestinal disorders) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 23 (27)
Alanine aminotransferase increased (Investigations) | 25 (53)
Alkaline phosphatase increased (Investigations) | 27 (50)
Allergic reaction (Immune system disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3)
Anemia (Blood and lymphatic system disorders) | 22 (54)
Anorexia (Metabolism and nutrition disorders) | 24 (32)
Anxiety (Psychiatric disorders) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 30 (66)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (7)
Bleeding (Epistaxis, Hematuria, Hematoma, Hemorrhoidal hemorrhage, Rectal hemorrhage) (Gastrointestinal disorders) | 5 (8)
Blood bilirubin increased (Investigations) | 14 (40)
Chest pain - cardiac (Cardiac disorders) | 2 (2)
Chills (General disorders) | 5 (5)
Confusion (Psychiatric disorders) | 5 (9)
Constipation (Gastrointestinal disorders) | 18 (24)
Cough (Respiratory, thoracic and mediastinal disorders) | 13 (16)
Dehydration (Metabolism and nutrition disorders) | 5 (7)
Depression (Psychiatric disorders) | 2 (2)
Diaphoresis (Skin and subcutaneous tissue disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 23 (50)
Dizziness (Nervous system disorders) | 8 (8)
Dry mouth (Gastrointestinal disorders) | 2 (2)
Dysgeusia (Nervous system disorders) | 2 (3)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9 (9)
Edema face (General disorders) | 2 (2)
Edema limbs (General disorders) | 8 (8)
Fall (Injury, poisoning and procedural complications) | 3 (6)
Fatigue (General disorders) | 34 (65)
Fever (General disorders) | 6 (6)
Flatulence (Gastrointestinal disorders) | 2 (2)
Flushing (Vascular disorders) | 2 (2)
Frequent urination (Investigations) | 2 (2)
Headache (Nervous system disorders) | 9 (9)
Hearing impaired (Ear and labyrinth disorders) | 2 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 28 (124)
Hyperkalemia (Metabolism and nutrition disorders) | 4 (4)
Hypertension (Vascular disorders) | 14 (21)
Hyperuricemia (Metabolism and nutrition disorders) | 3 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 12 (26)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (3)
Hypokalemia (Metabolism and nutrition disorders) | 6 (9)
Hypomagnesemia (Metabolism and nutrition disorders) | 7 (15)
Hyponatremia (Metabolism and nutrition disorders) | 17 (39)
Hypophosphatemia (Metabolism and nutrition disorders) | 25 (73)
Hypotension (Vascular disorders) | 2 (4)
Increased LDH (Investigations) | 3 (3)
INR increased (Investigations) | 3 (3)
Insomnia (Psychiatric disorders) | 11 (12)
Lipase increased (Investigations) | 16 (31)
Lymphocyte count decreased (Investigations) | 16 (47)
Memory impairment (Nervous system disorders) | 2 (2)
Mouth Sores (Gastrointestinal disorders) | 11 (18)
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 7 (8)
Nausea (Gastrointestinal disorders) | 27 (46)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Neutrophil count decreased (Investigations) | 14 (21)
Oral pain (Gastrointestinal disorders) | 2 (4)
Pain (General disorders) | 19 (42)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 13 (32)
Peripheral motor neuropathy (Nervous system disorders) | 2 (4)
Peripheral sensory neuropathy (Nervous system disorders) | 21 (35)
Platelet count decreased (Investigations) | 25 (59)
Proteinuria (Renal and urinary disorders) | 2 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (6)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 3 (6)
Rash (Skin and subcutaneous tissue disorders) | 17 (26)
Respiratory, thoracic and mediastinal disorders; other (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Serum amylase increased (Investigations) | 9 (20)
Thromboembolic event (Vascular disorders) | 2 (2)
Upper respiratory infection (Infections and infestations) | 5 (6)
Urinary tract infection (Infections and infestations) | 2 (3)
Urinary urgency (Renal and urinary disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 11 (15)
Weight loss (Investigations) | 8 (9)
White blood cell decreased (Investigations) | 9 (22)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-02-24): https://cdn.clinicaltrials.gov/large-docs/01/NCT01775501/Prot_SAP_000.pdf